CLINICAL TRIAL: NCT02520986
Title: Carbon Dioxide Laser Ablation Versus Electrocoagulation - a Prospective, Randomized Multicenter Trial Comparing Two Surgical Treatments in Women Undergoing Therapy for Condyloma Acuminata
Brief Title: Carbon Dioxide Laser vs. Electrocoagulation for the Therapy of Condyloma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zydolab - Institute of Cytology and Immune Cytochemistry (Other)
Collaborators: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Dr. med. Ziad Hilal, Dr. med. Ziad Hilal, Zydolab - Institute of Cytology and Immune Cytochemistry
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CONDYLOMA-1
Record Dates: First submitted 2015-08-04; First posted 2015-08-13 (Estimated); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Condylomata Acuminata
Keywords: Sexually transmitted disease; Genital Warts; Venereal Warts
MeSH Terms: conditions — Condylomata Acuminata; Sexually Transmitted Diseases | interventions — Electrocoagulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbon dioxide Laser ablation (Experimental): Excision of genital warts using a carbon dioxide laser, ie CO2 Laser
  Interventions: Device: Carbon dioxide Laser ablation
- Electrocoagulation (Active Comparator): Excision of genital warts using a superficial electrical coagulation mode, ie spray coagulation
  Interventions: Device: Electrocoagulation

INTERVENTIONS:
Device: Carbon dioxide Laser ablation — surgical Instrument to achieve excision of genital warts by a pulsed laser of 15 Watt voltage
  Arms: Carbon dioxide Laser ablation
Device: Electrocoagulation — surgical Instrument to achieve excision of genital warts by a deep tissue electrocoagulation of 80 Watt voltage
  Arms: Electrocoagulation

SUMMARY:
In a randomized clinical trial of 114 women undergoing Treatment for condyloma acuminata, two surgical methods, the carbon dioxide laser Ablation and the excision by electrocoagulation, will be compared. The primary outcome of the study is the cosmetic result judged by the Patient 6 weeks after Treatment using a 11-step visual analogue scale (VAS), secondary outcomes are intervention time, operative complications, subjects and users satisfaction, postoperative pain and recurrence of genital warts.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* women with anogenital affection of condyloma acuminata

Exclusion Criteria:

* significant language barrier
* pregnancy
* unwillingness to participate
* the use of blood thinner or known coagulation disorder
* the use of immunosuppressive medicament
* HIV-Infection
* malignant diseases
* local therapy within 8 weeks before Treatment
* wound healing disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Cosmetic result | 6 weeks
  Cosmetic result judged by the Patient 6 weeks after Treatment using a 11-step visual analogue scale (VAS)

SECONDARY OUTCOMES:
users satisfaction | 30 minutes
  surgeons will score their satisfaction concerning the used technique by using a 11-step visual analogue scale (VAS) within 30 minutes after surgery
Operation time | 20 minutes
  the time from the beginning of the Treatment until the end of the operation (the end of hemostatic interventions) will be measured in minutes
Postoperative pain | 5 hours
  patients will score their postoperative pain Level using a 11-step visual analogue scale (VAS) within 5 hours after surgery
Subjects satisfaction | 6 weeks
  Patients will score their Overall satisfaction by using a 11-step visual analogue scale (VAS) 6 weeks after Treatment
Recurrence of genital warts | 12 months
  an examination will be performed 12 months after surgery; Recurrence of genital warts will be determined if one or more Areas are infected by genital warts
Operative complications | 14 days
  Operative complications defined as necessity to intervene surgically up to 14 days postoperatively (number of patients with operative complications and type of complication)
Subjects satisfaction | 12 weeks
  Patients will score their Overall satisfaction by using a 11-step visual analogue scale (VAS) 12 weeks after Treatment
Cosmetic result | 12 weeks
  Cosmetic result judged by the Patient 12 weeks after Treatment using a 11-step visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Hilal, Dr. med., Principal Investigator — Zydolab - Institute of Cytology and Immune Cytochemistry
Locations (1):
- Department of Obstetrics and Gynecology of the Ruhr University Bochum, Herne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No